CLINICAL TRIAL: NCT06649526
Title: Comparison of Direct and Indirect Images of Two Different Video Laryngoscopes in Adult Airway Management
Brief Title: Comparison of Two Different Video Laryngoscopes
Status: Active, not recruiting | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Özlem Sezen, Associate Professor, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: Sezen
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Anesthesia
Keywords: video laryngoscopy; airway management; intubation
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group MC McGrath videolaryngoscope Group H Hugmed Videolaryngoscope: All patients will receive intravenous premedication with midazolam 0.03 mg/kg approximately 30 minutes before induction of anaesthesia. Preoperatively, standard monitoring included a 3-lead electrocardiogram (ECG) with continuous ST-segment analysis and assessment of peripheral oxygen saturation (SpO2) and intermittent non-invasive blood pressure. Following preoxygenation with 100% oxygen for three minutes, general anaesthesia would be induced with propofol (3mg/kg) a few minutes after injection of fentanyl (2µg/kg). Neuromuscular paralysis will be induced with rocuronium (0.5 mg/kg) in all patients.In group MC, direct and indirect Modified Cormack Lehane score and POGO score will be evaluated with McGrath videolaryngoscope.
  In Group H, direct and indirect Modified Cormack Lehane score and POGO score will be evaluated with Hugemed videolaryngoscope.
  Interventions: Other: endotracheal intubation with videolaryngoscope

INTERVENTIONS:
Other: endotracheal intubation with videolaryngoscope — The present study will compare the images of two different VLs with Macintosh blades (the McGrath videolaryngoscope and the Hugemed videolaryngoscope) in both indirect (screen images) and direct (images viewed through the mouth) laryngoscopy.

SUMMARY:
The aim of this study is to answer the question of whether direct laryngoscopy can be performed with videolaryngoscopes. How do the videos of the laryngoscopes provide images directly in laryngoscopy? Primary objective: To compare the images of Hugemed and Mcgrath videolarinygoscope in direct laryngoscopy and indirect laryngoscopy secondary objective: to compare the effects on haemodynamic response Participants :people who are not expected to have difficult intubation

DETAILED DESCRIPTION:
Direct and indirect images of hugemed and McGrath videolaryngoscope during intubation, haemodynamic responses, procedure time will be compared

ELIGIBILITY:
Inclusion Criteria:

To be between 18 -65 years old Mallampati score I-II Cormack-Lehane score I-II ASA physical status I-II who required endotracheal intubation for elective surgery

Exclusion criteria Pregnancy Mallampati score III-IV Cormack-Lehane score III-IV ASA physical score III-IV sternomental distance < 12.5 cm mandibular-hyoid distance < 6 cm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: After Ethics Committee approval and written informed consent were obtained, the study will be conducted with 70 patients aged 18-65 years and older of both sexes with American Society of Anaesthesiologists (ASA) physical status I-III. Patients will be divided into two groups by closed envelope method.
  McGrath video laryngoscope (MG) will be used in patients in group MC; Modified Cormack Lehane score and POGO score in direct laryngoscopic images and Modified Cormack Lehane score and POGO score in indirect laryngoscopic images of the patients will be evaluated and recorded and then orotracheal intubation will be performed.
  Hugemed videolaryngoscope (HG) will be used in patients in group H and orotracheal intubation will be performed after the Modified Cormack Lehane scores and POGO scores obtained from direct laryngoscopic and indirect laryngoscopic images of the patients are recorded.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of Direct and Indirect Images of Two Different Video Laryngoscopes in Adult Airway Management | 3 months
  Videolaryngoscopy (VL) is a frequently used method in airway management to improve the success of tracheal intubation in recent years. VLs have a miniature video camera at the tip of the blades which allows indirect visualisation of the glottis (1,2,3).
  The American Society of Anaesthesiologists (ASA) recommends that a VL should be available and used for all patients with a particularly difficult airway and for whom intubation is planned In recent years, a number of VLs have emerged that offer several advantages over direct laryngoscopy.It is aimed to compare direct and indirect images of mcgrath and hugemed videolaryngoscope.
Comparison of Direct and Indirect Images of Two Different Video Laryngoscopes in Adult Airway Management | 3 months
  The principal objective of this study was to undertake a comparative analysis of the images produced by two distinct VLs during direct and indirect laryngoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Kartal Dr. Lütfi Kirdar City Hospital Cevizli D-100 Güney Yanyol, No:47 Kartal Istanbul Turkey, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sezen O, Simsek T, Simsek AK, Arslan G, Saracoglu KT, Saracoglu A. Comparison of direct and indirect images and hemodynamic response of two different video laryngoscopes to tracheal intubation. BMC Anesthesiol. 2025 Feb 20;25(1):86. doi: 10.1186/s12871-025-02966-7. PMID 39979796